CLINICAL TRIAL: NCT04937868
Title: Developing a Decision Instrument to Guide Abdominal-pelvic CT Imaging of Blunt Trauma Patients
Acronym: NEXUS AP CT
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Brigham and Women's Hospital (Other); University of California, San Francisco (Other); Antelope Valley Hospital (Unknown); Stanford University (Other); UCSF - Fresno (Unknown); UC Davis (Unknown)
Responsible Party: Principal Investigator, William Mower, Professor of Emergency Medicine, David Geffen School of Medicine at UCLA, University of California, Los Angeles
Other Study IDs: 01APCT
Record Dates: First submitted 2021-05-24; First posted 2021-06-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Injury; Pelvic Fracture; Genital Hemorrhage; Lumbar Spine Injury; Hip Injuries; Liver Injury; Spleen Injury; Renal Injury; Diaphragm Injury; Aortic Rupture; Aortic Dissection; Bowel Disease; Vascular System Injuries; Sacral Fracture
Keywords: Blunt trauma; Abdominal injury; Pelvic injury; Spine injury; Genital injury; Vascular injury; Hip injury; Computed tomography; Decision instrument
MeSH Terms: conditions — Abdominal Injuries; Hip Fractures; Spinal Injuries; Hip Injuries; Aortic Rupture; Aortic Dissection; Intestinal Diseases; Vascular System Injuries; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blunt trauma patients undergoing abdominopelvic computed tomographic imaging: The study will be observational and not alter the care or management of blunt injury victims. Medical decisions will be made by treating physicians using current standards of care. Thus, to reduce the potential for bias, the study will seek to enroll all blunt injury victims who undergo A/P imaging as part of their ED trauma evaluation. This may include children, the elderly, all races, both sexes, and any other demographic or social groups that may present among blunt injury patients. An individual will become eligible for the study when the treating physician determines that A/P CT imaging is needed for their trauma evaluation. Inclusion or exclusion will not be based on age, gender, pregnancy or child-bearing potential, or racial/ethnic origin.
  There will be no exclusion criteria.
  Interventions: Other: There are no interventions associated with this study

INTERVENTIONS:
Other: There are no interventions associated with this study — This study is purely observational, there will be no interventions or changes in care related to patient inclusion in this study.

SUMMARY:
Unrecognized abdominal and pelvic injuries can result in catastrophic disability and death. Sporadic reports of "occult" injuries have generated concern, and physicians, fearing that they may miss such an injury, have adopted the practice of obtaining computed tomography on virtually all patients with significant blunt trauma. This practice exposes large numbers patients to dangerous radiation at considerable expense, while detecting injuries in a small minority of cases.

Existing data suggest that a limited number of criteria can reliably identify blunt injury victims who have "no risk" of abdominal or pelvic injuries, and hence no need for computed tomography (CT), without misidentifying any injured patient. It is estimated that nationwide implementation of such criteria could result in an annual reduction in radiographic charges of $75 million, and a significant decrease in radiation exposure and radiation induced malignancies.

This study seeks to determine whether "low risk" criteria can reliably identify patients who have sustained significant abdominal or pelvic injuries and safely decrease CT imaging of blunt trauma patients. This goal will be accomplished in the following manner:

All blunt trauma victims undergoing computed tomography of the abdomen/pelvis in the emergency department will undergo routine clinical evaluations prior to radiographic imaging. Based on these examinations, the presence or absence of specific clinical findings (i.e. abdominal/pelvic/flank pain, abdominal/pelvic/flank tenderness, bruising abrasions, distention, hip pain, hematuria, hypotension, tachycardia, low or falling hematocrit, intoxication, altered sensorium, distracting injury, positive FAST imaging, dangerous mechanism, abnormal x-ray imaging) will be recorded for each patient, as will the presence or absence of abdominal or pelvic injuries. The clinical findings will serve as potential imaging criteria. At the completion of the derivation portion of the study the criteria will be examined to find a subset that predicts injury with high sensitivity, while simultaneously excluding injury, and hence the need for imaging, in the remaining patients. These criteria will then be confirmed in a separate validation phase of the study.

The criteria will be considered to be reliable if the lower statistical confidence limit for the measured sensitivity exceeds 98.0%. Potential reductions in CT imaging will be estimated by determining the proportion of "low-risk" patients that do not have significant abdominal or pelvic injuries.

DETAILED DESCRIPTION:
RESEARCH STRATEGY

Significance

Injuries to the abdomen and pelvis can lead to significant morbidity and mortality in adult blunt trauma patients. Clinicians, concerned about abdominal and pelvic injuries, have increasingly utilized abdominal-pelvic (A/P) CT imaging of blunt trauma patients.

CT imaging is compelling because of its documented high sensitivity in detecting injuries, and has lead some to recommend "pan-scan" imaging, which includes head, neck, chest and A/P CT imaging, of all blunt trauma patients. However, well-designed comparative trials have repeatedly failed to demonstrate improved patient outcomes thorough the use of "pan-scanning". It is hard to justify routine imaging if there is no benefit, particularly since A/P CT imaging is expensive and exposes patients to ionizing radiation and risk of lethal malignant transformation. As a consequence, recent recommendations emphasize the use of selective imaging in assessing most trauma patients.

At the present time, there are no definite recommendations to guide selective A/P CT imaging of blunt trauma patients. In current practice, imaging decisions are typically based on clinical judgment, which suffers from poor specificity and substantial variability, making it an imprecise and unreliable tool. A rigorously develop decision instrument could provide substantial benefit in guiding selective A/P CT imaging.

A decrease in CT utilization by as little as 10% would translate to substantial, direct, long-term benefits. There were approximately 1.5 million blunt trauma activation visits at the 1,632 adult trauma centers in the United States in 2015. Nearly half of these patients underwent abdominal-pelvic CT imaging, implying that nation-wide approximately 750,000 blunt trauma patients undergo A/P CT imaging each year. If a decision instrument could allow clinicians to safely forego at least 10% of these CTs, up to 75,000 CTs could be eliminated annually in the U.S. This reduction would provide cost and resource savings, reduced radiation exposure and iatrogenic cancers in the young vulnerable trauma population, and facilitate more efficient trauma evaluations, translating to shorter ED length of stay.

Approach

Investigators will employ the classic design strategy described by Stiell in developing the decision instrument. The development process includes separate derivation and validation phases. The clinical criteria identified in the derivation phase will form the basis of the instrument, with "high-risk" classification assigned to patients exhibiting one or more of the criteria, and "low-risk" classification assigned to patients who exhibit none of the criteria. Investigators will then conduct a separate validation assessment to determine whether the instrument retains optimal performance among a new cohort of patients. The validation phase will focus on ensuring that the final instrument has the high sensitivity and negative predictive value (NPV) needed to ensure its safe application, while retaining the highest possible specificity (and potential to decrease imaging).

The primary goal of the study will be to develop an instrument that reliably identifies patients who have injuries of major clinical significance that are evident on A/P CT imaging. The injuries of interest in this goal include injuries that require intervention, as well as any injuries to the aorta (including those not requiring intervention), and select injuries to the spine.

The secondary goal of the study will be to develop a tool that reliably identifies patients who have injuries of major or minor clinical significance. The injuries of interest related to this goal include injuries that require intervention, injuries that merit clinical observation, any injuries to the aorta, and select injuries to the spine.

To be clinically reliable, the DI must exhibit a sensitivity and negative predictive value of 98% or greater. At this level of precision, the risk of unfavorable outcomes due to missed injuries is equivalent to the risk of lethal malignant transformation from the radiation exposure associated with increased imaging. Validating a 95% lower confidence bound of 98.0% for a measured NPV of 100.0% requires evaluations on 183 patients assigned "low risk" status by the instrument. Similar validation of the sensitivity requires evaluations on 183 patients who have sustained injuries of major clinical significance. Because "low risk" patients are more prevalent than those sustaining major injuries, the ultimate sample estimate is driven by the need to enroll 183 patients who have sustained major A/P injuries.

Protocol

Phase I - Derivation

Clinicians will assess the presence or absence of each of the candidate criteria for each imaged patient during their initial emergency department evaluation. These assessments will be recorded prior to initiating CT imaging.

The injury status of each patient will be based on final radiologic interpretation of the initial A/P CT imaging obtained in the ED. Investigators require that relevant injuries be evident on CT imaging because the risk classification assigned by the instrument is immaterial if an injury is not visible on CT imaging. Injuries will be further classified as being of major, minor, or insignificant concern based on review of the patients care during their index visit.

The three level injury classification reflects the fact that many clinicians are comfortable in missing minor injuries provided that all injuries requiring intervention are identified, while other clinicians are uncomfortable using tools that occasionally miss minor injuries that require no intervention, and seek to identify all injuries regardless of their clinical significance.

To accommodate these perspectives, investigators will employ identical techniques to develop a two separate decision instruments. The first, and primary goal of the study, is to develop an instrument that identifies all injuries requiring intervention, while a second goal is to create an instrument that identifies all significant injuries, whether they require intervention or not.

Investigators will employ binary recursive partitioning to derive the decision instruments. The primary instrument must exhibit a sensitivity and negative predictive value greater than 98.0% in detecting and excluding major injuries. The second instrument must exhibit similar sensitivity and NPV in detecting and excluding major and minor injuries.

Phase II - Validation

In the second phase of the study, investigators will apply the instruments to a new cohort of blunt trauma patients to assess their performance and determine whether they retain sufficient sensitivity to support their use as A/P CT decision tools.

Clinicians will again document the presence or absence of criteria during their initial emergency department evaluations, and record their impressions prior to imaging. Investigators will base the presence or absence of injury on the final radiologic interpretation of the initial A/P CT imaging obtained in the ED. Injuries will be further classified as being of major, minor, or insignificant concern based on review of the patients care during their index visit.

The primary outcome will be the sensitivity of the instrument in classifying as "high-risk" all patients harboring injuries of major importance. Investigators will also calculate the NPV, specificity, and count the number of "low-risk" patients for whom imaging might have been safely omitted had the decision instrument been implemented.

The secondary outcome will be to perform a similar analysis focused on identifying patients with injuries major or minor clinical significance, and will measure the sensitivity, NPV, specificity, and potential to reduce imaging using this additional version of the instrument.

Data Collection

Criteria assessments.

Physicians will assess the status of the individual criteria during their initial emergency department evaluations and prior to ordering CT imaging. Investigators will record demographic information for each patient, along with the clinician assessments of the presence or absence of potential predictor variables. The potential predictor variables include abdominal pain or tenderness, flank pain or tenderness, pelvic pain or tenderness, hip or iliac pain or tenderness, midline lumbar spine or sacral pain, abnormal alertness, evidence of intoxication, distracting painful injury, and hypotension. Investigators will also record historical information and emergency department vital signs measurements.

Data collection during the validation phase will follow a similar process, but will be limited to demographic information and the criteria that compose the decision instruments.

Patient outcomes.

The presence of significant major or minor injuries will be based on final radiologic interpretation of the initial CT imaging obtained in the ED. The classification into major or minor status will be based on review of the patients care during their index visit to determine whether the patient underwent any interventional procedures.

All injury assessments will be completed by trained investigators blinded to criteria assessments and final classification by the decision instrument. Investigators require that relevant injuries for the study must be evident on CT imaging because risk classification assigned by the instrument is immaterial if an injury is not visible on CT imaging.

Injuries of major clinical significance consist of all abdominal and pelvic injuries requiring intervention, as well as any injury to the aorta, and any injury to the spine involving instability or neurological compromise. Injuries that require only observation, but no intervention, will be considered clinically minor, provided they do not involve the aorta or spine, while injuries that required neither intervention nor observation, and that do not involve the aorta or spine will be considered insignificant.

Formulation of the optimal A/P CT decision instrument.

Investigators will treat each individual criterion as a dichotomous variable. For analytic purposes in the derivation phase, each variable will be considered negative (normal) unless it can be assessed and found to be abnormal. Thus, variables that cannot be measured in an individual patient (such as coagulopathy in an unconscious individual) will be documented as "unable to assess" and treated statistically as negative. This will ensure that the derivation process is based on observed assessments and is as robust as possible. Investigators will use the individual criteria to construct the nodal points of the recursive partitions.

Investigators will employ binary recursive partitioning to identify a combination of candidate criteria that predicts significant abdominal-pelvic injuries with > 98.0% sensitivity, excludes significant injuries with > 98.0% NPV, and retains the greatest specificity. Sensitivity will be used as the outcome measure for constructing the partitions. Investigators will terminate the partitioning under the following circumstances: 1) partitioning produces an instrument exhibiting a sensitivity of 100.0%, 2) partitioning exhausts all patients without developing a sufficiently sensitive rule, 3) partitioning exhausts all variables (criteria) without identifying a sufficiently sensitive rule. Circumstance I will confirm the hypothesis driving the first specific aim. Circumstance 2 and 3 may confirm the first hypothesis, provided the lower confidence limit of for the sensitivity of the resultant rule exceeds 98.0%, otherwise these circumstances will be interpreted to refute the first hypothesis.

Investigators will create two distinct decision instruments. The first, and primary instrument will focus on identifying only those patients having injuries of major clinical significance. Investigators will also develop a second instrument that identifies patients having injuries of either major or minor significance.

Validation of the A/P CT decision instrument.

The validation phase will again treat each individual criterion as a dichotomous variable. Each variable will be considered negative (normal) only if it is assessed and found to be normal. Variables that cannot be measured in an individual patient (i.e. coagulopathy in an unconscious individual) will be documented as "un-assessable" and treated statistically as positive. This ensures that patients will be assigned low-risk status only if all criteria are adequately assessed and found to be negative. Patients will be excluded from low-risk classification (and assigned high-risk status) if they have one or more positive or un-assessed criteria. This requirement ensures patients are not assigned low-risk status on the basis of an inadequate assessment.

Using the final risk assignments and patient outcomes, investigators will assign each case to one of the following four categories: 1 - true-positive status (injured patients classified as "high-risk" by the DI); 2 - false-negative status (injured patients classified as "low-risk" by the DI); 3 - false-positive status (uninjured patients classified as "high-risk" by the DI); and 4 - true-negative status (uninjured patients classified as "low-risk" by the DI). Investigators will employ these values to calculate point measures and 95 percent confidence intervals for sensitivity, NPV and specificity of the decision instrument. Investigators will consider the instrument to be validated if the lower 95% confidence interval for its measured sensitivity exceeds 98.0%.

Assessing the potential to decrease A/P CT imaging.

Investigators must assess whether application of the tool to blunt trauma patients actually has the potential to decrease A/P CT imaging. Because of the tool's inherent sensitivity, "low risk" patients will be free of injury and receive no benefit from imaging. They are ideal candidates to exclude from imaging. Thus, measuring the proportion of "low-risk" patients will provide the investigators with an estimate of potential imaging reductions. Reductions in charges and radiation exposure will be determined by respectively summing radiographic charges and life-time decreases in radiation morbidity and mortality for all "no risk" cases.

ELIGIBILITY:
Inclusion Criteria:

Blunt trauma patients who undergo abdominal-pelvic CT imaging during their initial trauma evaluation in the emergency department.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All blunt injury victims who undergo A/P imaging as part of their ED trauma evaluation. This may include children, the elderly, all races, both sexes, and any other demographic or social groups that may present among blunt injury patients. An individual will become eligible for the study when the treating physician determines that A/P CT imaging is needed for their trauma evaluation. Inclusion or exclusion will not be based on age, gender, pregnancy or child-bearing potential, or racial/ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Detection of injuries of major clinical significance | Initial abdominal-pelvic imaging on the 1 day of presentation.
  Injuries of major clinical significance consist of all abdominal and pelvic injuries requiring intervention, as well as any injury to the aorta, and any injury to the spine involving instability or neurological compromise.
Detection of injuries of major or minor clinical importance | Initial abdominal-pelvic imaging on the 1 day of presentation.
  Detect the presences of all abdominal and pelvic injuries requiring intervention or observation, including all abdominal and pelvic injuries requiring intervention, as well as any injury to the aorta, and any injury to the spine involving instability or neurological compromise.

CONTACTS AND LOCATIONS:
Overall Officials: William R Mower, MD, PhD, Study Director — University of California, Los Angeles
Locations (1):
- Ronald Reagan Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study we plan to make a de-identified version of our database that contains individual patient demographic information, physician assessments and outcome/injury assessments, available in a public repository.
Supporting Information: Study Protocol, SAP
Time Frame: We anticipate data will become available in the next two to four years, and will be available for a period of seven years.
Access Criteria: To be determined

REFERENCES:
- [Background] Sugrue M, Caldwell E, D'Amours S, Crozier J, Wyllie P, Flabouris A, Sheridan M, Jalaludin B. Time for a change in injury and trauma care delivery: a trauma death review analysis. ANZ J Surg. 2008 Nov;78(11):949-54. doi: 10.1111/j.1445-2197.2008.04711.x. PMID 18959692
- [Background] Hilty MP, Behrendt I, Benneker LM, Martinolli L, Stoupis C, Buggy DJ, Zimmermann H, Exadaktylos AK. Pelvic radiography in ATLS algorithms: A diminishing role? World J Emerg Surg. 2008 Mar 4;3:11. doi: 10.1186/1749-7922-3-11. PMID 18318904
- [Background] Kortbeek JB, Al Turki SA, Ali J, Antoine JA, Bouillon B, Brasel K, Brenneman F, Brink PR, Brohi K, Burris D, Burton RA, Chapleau W, Cioffi W, Collet e Silva Fde S, Cooper A, Cortes JA, Eskesen V, Fildes J, Gautam S, Gruen RL, Gross R, Hansen KS, Henny W, Hollands MJ, Hunt RC, Jover Navalon JM, Kaufmann CR, Knudson P, Koestner A, Kosir R, Larsen CF, Livaudais W, Luchette F, Mao P, McVicker JH, Meredith JW, Mock C, Mori ND, Morrow C, Parks SN, Pereira PM, Pogetti RS, Ravn J, Rhee P, Salomone JP, Schipper IB, Schoettker P, Schreiber MA, Smith RS, Svendsen LB, Taha W, van Wijngaarden-Stephens M, Varga E, Voiglio EJ, Williams D, Winchell RJ, Winter R. Advanced trauma life support, 8th edition, the evidence for change. J Trauma. 2008 Jun;64(6):1638-50. doi: 10.1097/TA.0b013e3181744b03. PMID 18545134
- [Background] Raja AS, Mortele KJ, Hanson R, Sodickson AD, Zane R, Khorasani R. Abdominal imaging utilization in the emergency department: trends over two decades. Int J Emerg Med. 2011 Apr 27;4:19. doi: 10.1186/1865-1380-4-19. PMID 21584210
- [Background] Lee J, Kirschner J, Pawa S, Wiener DE, Newman DH, Shah K. Computed tomography use in the adult emergency department of an academic urban hospital from 2001 to 2007. Ann Emerg Med. 2010 Dec;56(6):591-6. doi: 10.1016/j.annemergmed.2010.05.027. PMID 20619935
- [Background] Obaid AK, Barleben A, Porral D, Lush S, Cinat M. Utility of plain film pelvic radiographs in blunt trauma patients in the emergency department. Am Surg. 2006 Oct;72(10):951-4. doi: 10.1177/000313480607201025. PMID 17058743
- [Background] Deunk J, Brink M, Dekker HM, Kool DR, Blickman JG, van Vugt AB, Edwards MJ. Predictors for the selection of patients for abdominal CT after blunt trauma: a proposal for a diagnostic algorithm. Ann Surg. 2010 Mar;251(3):512-20. doi: 10.1097/SLA.0b013e3181cfd342. PMID 20083993
- [Background] Holmes JF, Wisner DH, McGahan JP, Mower WR, Kuppermann N. Clinical prediction rules for identifying adults at very low risk for intra-abdominal injuries after blunt trauma. Ann Emerg Med. 2009 Oct;54(4):575-84. doi: 10.1016/j.annemergmed.2009.04.007. Epub 2009 May 19. PMID 19457583
- [Background] Duane TM, Tan BB, Golay D, Cole FJ Jr, Weireter LJ Jr, Britt LD. Blunt trauma and the role of routine pelvic radiographs: a prospective analysis. J Trauma. 2002 Sep;53(3):463-8. doi: 10.1097/01.TA.0000025381.48450.6C. PMID 12352481
- [Background] Holmes JF, Sokolove PE, Brant WE, Palchak MJ, Vance CW, Owings JT, Kuppermann N. Identification of children with intra-abdominal injuries after blunt trauma. Ann Emerg Med. 2002 May;39(5):500-9. doi: 10.1067/mem.2002.122900. PMID 11973557
- [Background] Rose JS, Richards JR, Battistella F, Bair AE, McGahan JP, Kuppermann N. The fast is positive, now what? Derivation of a clinical decision rule to determine the need for therapeutic laparotomy in adults with blunt torso trauma and a positive trauma ultrasound. J Emerg Med. 2005 Jul;29(1):15-21. doi: 10.1016/j.jemermed.2005.01.004. PMID 15961002
- [Background] Ali J, Ahmadi KA, Williams JI. Predictors of laparotomy and mortality in polytrauma patients with pelvic fractures. Can J Surg. 2009 Aug;52(4):271-276. PMID 19680510
- [Background] Davis JW, Mackersie RC, Holbrook TL, Hoyt DB. Base deficit as an indicator of significant abdominal injury. Ann Emerg Med. 1991 Aug;20(8):842-4. doi: 10.1016/s0196-0644(05)81423-4. PMID 1854065
- [Background] Mackersie RC, Tiwary AD, Shackford SR, Hoyt DB. Intra-abdominal injury following blunt trauma. Identifying the high-risk patient using objective risk factors. Arch Surg. 1989 Jul;124(7):809-13. doi: 10.1001/archsurg.1989.01410070063013. PMID 2742481
- [Background] Nishijima DK, Simel DL, Wisner DH, Holmes JF. Does this adult patient have a blunt intra-abdominal injury? JAMA. 2012 Apr 11;307(14):1517-27. doi: 10.1001/jama.2012.422. PMID 22496266
- [Background] Richards JR, Derlet RW. Computed tomography and blunt abdominal injury: patient selection based on examination, haematocrit and haematuria. Injury. 1997 Apr;28(3):181-5. doi: 10.1016/s0020-1383(96)00187-8. PMID 9274733
- [Background] Wuthisuthimethawee P. Predictive factors for a FAST-positive and a therapeutic laparotomy in blunt abdominal injuries at the emergency room. J Med Assoc Thai. 2012 Mar;95(3):337-41. PMID 22550831
- [Background] Lagisetty J, Slovis T, Thomas R, Knazik S, Stankovic C. Are routine pelvic radiographs in major pediatric blunt trauma necessary? Pediatr Radiol. 2012 Jul;42(7):853-8. doi: 10.1007/s00247-011-2341-7. Epub 2012 Jan 14. PMID 22246414
- [Background] Yoong S, Kothari R, Brooks A. Assessment of sensitivity of whole body CT for major trauma. Eur J Trauma Emerg Surg. 2019 Jun;45(3):489-492. doi: 10.1007/s00068-018-0926-7. Epub 2018 Mar 8. PMID 29520416
- [Background] Benjamin E, Cho J, Recinos G, Dilektasli E, Lam L, Brunner J, Inaba K, Demetriades D. Negative computed tomography can safely rule out clinically significant intra-abdominal injury in the asymptomatic patient after blunt trauma: Prospective evaluation of 1193 patients. J Trauma Acute Care Surg. 2018 Jan;84(1):128-132. doi: 10.1097/TA.0000000000001705. PMID 28930944
- [Background] Huber-Wagner S, Lefering R, Qvick LM, Korner M, Kay MV, Pfeifer KJ, Reiser M, Mutschler W, Kanz KG; Working Group on Polytrauma of the German Trauma Society. Effect of whole-body CT during trauma resuscitation on survival: a retrospective, multicentre study. Lancet. 2009 Apr 25;373(9673):1455-61. doi: 10.1016/S0140-6736(09)60232-4. Epub 2009 Mar 25. PMID 19321199
- [Background] Huber-Wagner S, Biberthaler P, Haberle S, Wierer M, Dobritz M, Rummeny E, van Griensven M, Kanz KG, Lefering R; TraumaRegister DGU. Whole-body CT in haemodynamically unstable severely injured patients--a retrospective, multicentre study. PLoS One. 2013 Jul 24;8(7):e68880. doi: 10.1371/journal.pone.0068880. Print 2013. PMID 23894365
- [Background] Wurmb TE, Quaisser C, Balling H, Kredel M, Muellenbach R, Kenn W, Roewer N, Brederlau J. Whole-body multislice computed tomography (MSCT) improves trauma care in patients requiring surgery after multiple trauma. Emerg Med J. 2011 Apr;28(4):300-4. doi: 10.1136/emj.2009.082164. Epub 2010 Jul 20. PMID 20659885
- [Background] Yeguiayan JM, Yap A, Freysz M, Garrigue D, Jacquot C, Martin C, Binquet C, Riou B, Bonithon-Kopp C; FIRST Study Group. Impact of whole-body computed tomography on mortality and surgical management of severe blunt trauma. Crit Care. 2012 Jun 11;16(3):R101. doi: 10.1186/cc11375. PMID 22687140
- [Background] Wada D, Nakamori Y, Yamakawa K, Yoshikawa Y, Kiguchi T, Tasaki O, Ogura H, Kuwagata Y, Shimazu T, Hamasaki T, Fujimi S. Impact on survival of whole-body computed tomography before emergency bleeding control in patients with severe blunt trauma. Crit Care. 2013 Aug 27;17(4):R178. doi: 10.1186/cc12861. PMID 24025196
- [Background] Sierink JC, Saltzherr TP, Beenen LF, Luitse JS, Hollmann MW, Reitsma JB, Edwards MJ, Hohmann J, Beuker BJ, Patka P, Suliburk JW, Dijkgraaf MG, Goslings JC; REACT-2 study group. A multicenter, randomized controlled trial of immediate total-body CT scanning in trauma patients (REACT-2). BMC Emerg Med. 2012 Mar 30;12:4. doi: 10.1186/1471-227X-12-4. PMID 22458247
- [Background] Sierink JC, Treskes K, Edwards MJ, Beuker BJ, den Hartog D, Hohmann J, Dijkgraaf MG, Luitse JS, Beenen LF, Hollmann MW, Goslings JC; REACT-2 study group. Immediate total-body CT scanning versus conventional imaging and selective CT scanning in patients with severe trauma (REACT-2): a randomised controlled trial. Lancet. 2016 Aug 13;388(10045):673-83. doi: 10.1016/S0140-6736(16)30932-1. Epub 2016 Jun 28. PMID 27371185
- [Background] Moussavi N, Ghani H, Davoodabadi A, Atoof F, Moravveji A, Saidfar S, Talari H. Routine versus selective chest and abdominopelvic CT-scan in conscious blunt trauma patients: a randomized controlled study. Eur J Trauma Emerg Surg. 2018 Feb;44(1):9-14. doi: 10.1007/s00068-017-0842-2. Epub 2017 Sep 25. PMID 28948295
- [Background] Palm HG, Kulla M, Wettberg M, Lefering R, Friemert B, Lang P; TraumaRegistrer DGU(R). Changes in trauma management following the implementation of the whole-body computed tomography: a retrospective multi-centre study based on the trauma registry of the German Trauma Society (TraumaRegister DGU(R)). Eur J Trauma Emerg Surg. 2018 Oct;44(5):759-766. doi: 10.1007/s00068-017-0870-y. Epub 2017 Nov 3. PMID 29101416
- [Background] Long B, April MD, Summers S, Koyfman A. Whole body CT versus selective radiological imaging strategy in trauma: an evidence-based clinical review. Am J Emerg Med. 2017 Sep;35(9):1356-1362. doi: 10.1016/j.ajem.2017.03.048. Epub 2017 Mar 21. PMID 28366287
- [Background] Inaba K, Branco BC, Lim G, Russell K, Teixeira PG, Lee K, Talving P, Reddy S, Demetriades D. The increasing burden of radiation exposure in the management of trauma patients. J Trauma. 2011 Jun;70(6):1366-70. doi: 10.1097/TA.0b013e3181ebb4d4. PMID 20962680
- [Background] Kendall JL, Kestler AM, Whitaker KT, Adkisson MM, Haukoos JS. Blunt abdominal trauma patients are at very low risk for intra-abdominal injury after emergency department observation. West J Emerg Med. 2011 Nov;12(4):496-504. doi: 10.5811/westjem.2010.11.2016. PMID 22224146
- [Background] Sise MJ, Kahl JE, Calvo RY, Sise CB, Morgan JA, Shackford SR, Shackford MC, Bandle J, Peck KA, Schechter MS. Back to the future: reducing reliance on torso computed tomography in the initial evaluation of blunt trauma. J Trauma Acute Care Surg. 2013 Jan;74(1):92-7; discussion 97-9. doi: 10.1097/TA.0b013e3182788f6f. PMID 23271082
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] Laupacis A, Sekar N, Stiell IG. Clinical prediction rules. A review and suggested modifications of methodological standards. JAMA. 1997 Feb 12;277(6):488-94. PMID 9020274
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Melnick ER, Keegan J, Taylor RA. Redefining Overuse to Include Costs: A Decision Analysis for Computed Tomography in Minor Head Injury. Jt Comm J Qual Patient Saf. 2015 Jul;41(7):313-22. doi: 10.1016/s1553-7250(15)41041-4. PMID 26108124
- [Background] Tillou A, Gupta M, Baraff LJ, Schriger DL, Hoffman JR, Hiatt JR, Cryer HM. Is the use of pan-computed tomography for blunt trauma justified? A prospective evaluation. J Trauma. 2009 Oct;67(4):779-87. doi: 10.1097/TA.0b013e3181b5f2eb. PMID 19820586
- [Background] Gupta M, Schriger DL, Hiatt JR, Cryer HG, Tillou A, Hoffman JR, Baraff LJ. Selective use of computed tomography compared with routine whole body imaging in patients with blunt trauma. Ann Emerg Med. 2011 Nov;58(5):407-16.e15. doi: 10.1016/j.annemergmed.2011.06.003. Epub 2011 Sep 3. PMID 21890237
- [Derived] Raja AS, Rodriguez RM, Gupta M, Isaacs ED, Kornblith LZ, Prabhakar A, Saillant N, Schmit PJ, Wei SH, Mower WR. Developing a decision instrument to guide abdominal-pelvic imaging of blunt trauma patients: Methodology and protocol of the NEXUS abdominal-pelvic imaging study. PLoS One. 2022 Jul 25;17(7):e0271070. doi: 10.1371/journal.pone.0271070. eCollection 2022. PMID 35877687